CLINICAL TRIAL: NCT06947564
Title: Angiography-derived Index of Microcirculatory Resistance Predicts Microvascular Obstruction and Infarct Size in Patients With ST-segment-elevation Myocardial Infarction
Brief Title: AccuIMR Predicts Microvascular Obstruction and Infarct Size in STEMI Patients
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Early MYO IMR-CMR
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; STEMI - ST Elevation Myocardial Infarction; Microvascular Coronary Artery Disease
Keywords: AccuIMR, CMR, infarct size
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI patients underwent CMR: STEMI patients who underwent PCI within 12 hours of symptom onset.
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: CMR — Coronary microvascular function was assessed using contrast-enhanced CMR after PCI.

SUMMARY:
In this study, we aimed to investigate the clinical significance of the angiography-based IMR calculation method (AccuIMR) and its prognostic assessment capability by evaluating the concordance or discordance between AccuIMR values and cardiac magnetic resonance (CMR) results.

ELIGIBILITY:
Inclusion Criteria:

* (1) STEMI patients who underwent PCI within 12 hours of symptom onset.
* (2) coronary microvascular function was assessed using contrast-enhanced CMR after PCI.

Exclusion Criteria:

* (1) Suboptimal coronary angiographic images, including inadequate contrast opacification, unsatisfactory projection view, and severe overlap or distortion of the target vessel.
* (2) Lacking two angiographic projections separated by at least 25° apart post-PCI.
* (3) Inadequate CMR image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients who underwent PCI within 12 hours of symptom onset, and coronary microvascular function was assessed using contrast-enhanced CMR after PCI.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
CMR | CMR was performed at a median of 5 days post-reperfusion.
  Contrast-enhanced CMR was performed on a 3.0-T scanner (Achieva TX, Philips Healthcare, Best, The Netherlands) . All sequences were acquired during breath-hold with a field of view at 350 × 350 mm2. Two experienced readers, blinded to clinical data, evaluated the CMR results using validated software (QMass MR 7.5, Medis, Leiden, The Netherlands). The acquired images were utilized to assess ventricular parameters and calculate the left ventricular ejection fraction (LVEF).

SECONDARY OUTCOMES:
LDL-C, mmol/L | Blood samples were collected after a 12-hour fast in the second day post-PCI.
  Low-density cholesterol (LDL-C) is the cholesterol in low-density lipoprotein (LDL), which reflects how much LDL is present.
HbA1c, % | Blood samples were collected after a 12-hour fast in the second day post-PCI.
  Hemoglobin a1c (HbA1c) is the combination of hemoglobin and blood sugar. Its concentration in the blood is stable and is not affected by short-term blood sugar concentrations. Hemoglobin A1C has obvious clinical value in the diagnosis of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD, PhD, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Frampton J, Devries JT, Welch TD, Gersh BJ. Modern Management of ST-Segment Elevation Myocardial Infarction. Curr Probl Cardiol. 2020 Mar;45(3):100393. doi: 10.1016/j.cpcardiol.2018.08.005. Epub 2018 Sep 14. PMID 30660333
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, Schnittger I, Lee DP, Vagelos RH, Fitzgerald PJ, Yock PG, Yeung AC. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5. doi: 10.1016/j.jacc.2007.08.062. PMID 18237685
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Scarsini R, Kotronias RA, Della Mora F, Portolan L, Andreaggi S, Benenati S, Marin F, Sgreva S, Comuzzi A, Butturini C, Pesarini G, Tavella D, Channon KM, Garcia Garcia HM, Ribichini F, Banning AP, De Maria GL. Angiography-Derived Index of Microcirculatory Resistance to Define the Risk of Early Discharge in STEMI. Circ Cardiovasc Interv. 2024 Mar;17(3):e013556. doi: 10.1161/CIRCINTERVENTIONS.123.013556. Epub 2024 Feb 20. PMID 38375667
- [Background] Jiang J, Li C, Hu Y, Li C, He J, Leng X, Xiang J, Ge J, Wang J. A novel CFD-based computed index of microcirculatory resistance (IMR) derived from coronary angiography to assess coronary microcirculation. Comput Methods Programs Biomed. 2022 Jun;221:106897. doi: 10.1016/j.cmpb.2022.106897. Epub 2022 May 18. PMID 35636354
- [Background] Zhang Y, Pu J, Niu T, Fang J, Chen D, Yidilisi A, Zheng Y, Lu J, Hu Y, Koo BK, Xiang J, Wang J, Jiang J. Prognostic Value of Coronary Angiography-Derived Index of Microcirculatory Resistance in Non-ST-Segment Elevation Myocardial Infarction Patients. JACC Cardiovasc Interv. 2024 Aug 26;17(16):1874-1886. doi: 10.1016/j.jcin.2024.04.048. Epub 2024 Aug 7. PMID 39115479
- [Background] Yidilisi A, Chen D, Zhang Y, Pu J, Niu T, Hu Y, Fang J, Gong Q, Zheng Y, Huang J, Xiang J, Wang Y, Wang J, Jiang J. Coronary Angiography-Derived Index of Microcirculatory Resistance Predicts Outcome in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2024 May;17(5):e013899. doi: 10.1161/CIRCINTERVENTIONS.123.013899. Epub 2024 Apr 25. No abstract available. PMID 38660822
- [Background] Fan Y, Li C, Hu Y, Hu X, Wang S, He J, Leng X, Xiang J, Lu Z. Angiography-based index of microcirculatory resistance (AccuIMR) for the assessment of microvascular dysfunction in acute coronary syndrome and chronic coronary syndrome. Quant Imaging Med Surg. 2023 Jun 1;13(6):3556-3568. doi: 10.21037/qims-22-961. Epub 2023 Apr 17. PMID 37284070
- [Background] Symons R, Pontone G, Schwitter J, Francone M, Iglesias JF, Barison A, Zalewski J, de Luca L, Degrauwe S, Claus P, Guglielmo M, Nessler J, Carbone I, Ferro G, Durak M, Magistrelli P, Lo Presti A, Aquaro GD, Eeckhout E, Roguelov C, Andreini D, Vogt P, Guaricci AI, Mushtaq S, Lorenzoni V, Muller O, Desmet W, Agati L, Janssens S, Bogaert J, Masci PG. Long-Term Incremental Prognostic Value of Cardiovascular Magnetic Resonance After ST-Segment Elevation Myocardial Infarction: A Study of the Collaborative Registry on CMR in STEMI. JACC Cardiovasc Imaging. 2018 Jun;11(6):813-825. doi: 10.1016/j.jcmg.2017.05.023. Epub 2017 Aug 16. PMID 28823746
- [Background] De Maria GL, Alkhalil M, Wolfrum M, Fahrni G, Borlotti A, Gaughran L, Dawkins S, Langrish JP, Lucking AJ, Choudhury RP, Porto I, Crea F, Dall'Armellina E, Channon KM, Kharbanda RK, Banning AP. Index of Microcirculatory Resistance as a Tool to Characterize Microvascular Obstruction and to Predict Infarct Size Regression in Patients With STEMI Undergoing Primary PCI. JACC Cardiovasc Imaging. 2019 May;12(5):837-848. doi: 10.1016/j.jcmg.2018.02.018. Epub 2018 Apr 18. PMID 29680355
- [Background] Qi Y, Gu R, Xu J, Kang L, Liu Y, Wang L, Chen J, Zhang J, Wang K. Index of microcirculatory resistance predicts long term cardiac systolic function in patients with STEMI undergoing primary PCI. BMC Cardiovasc Disord. 2021 Feb 2;21(1):66. doi: 10.1186/s12872-021-01887-w. PMID 33530931